

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH WITH OPTIONAL PROCEDURES

Phase I/II Trial Immunotherapy with Durvalumab and Tremelimumab with Continuous or Intermittent MEK Inhibitor Selumetinib in NSCLC 2017-0888

| Study Chair: | Don L. Gibbons | | |
|--------------------|----------------|------------------|---|
| Participant's Name | Medic | al Record Number | _ |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to learn if adding selumetinib to durvalumab and tremelimumab can help to control non-small cell lung cancer (NSCLC). Researchers will also study 2 different dosing schedules of selumetinib.

**This is an investigational study.** Selumetinib and tremelimumab are not FDA approved or commercially available. Durvalumab is FDA approved for urothelial carcinoma. All the drugs are currently being used for research purposes. The study doctor can explain how the study drugs are designed to work.

The study doctor can explain how the study drugs are designed to work.

The study drugs may help control the disease. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects (such as skin rash or inflammation), potential expenses, and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may receive selumetinib and durvalumab for as long as the doctor thinks is in your best interest. You may receive tremelimumab for up to 4 cycles. If you complete the 4 cycles of treatment with selumetinib, durvalumab, and tremelimumab and the disease later gets worse while you are receiving selumetinib and durvalumab, you may be able to restart treatment with all 3 drugs for an additional 4 cycles. This may only be done 1 time and this possibility will be discussed with you.

Durvalumab, selumetinib, and tremelimumab will be provided at no cost to you during the study. You and/or your insurance provider will be responsible for the cost of any supportive drugs that you receive.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive FDA approved drug dabrafenib plus trametinib, if you have BRAF V600E mutation. You also may choose to have treatment with a single anti-PD-1/PD-L1 drug, if the disease got worse after platinum-based chemotherapy. You may also choose to have a combination of ramucirumab plus docetaxel or a platinum-doublet chemotherapy, if you have already had pembrolizumab as a single agent for first-line treatment. You may choose to receive other chemotherapy drugs or investigational therapy if available. The study doctor will discuss with you the possible risks and benefits of these treatments. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

## **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. You will have screening tests to help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an eye exam by an eye doctor.
- You will have an EKG and an echocardiogram (ECHO) or MUGA scan to check your heart function.
- You will have either a CT scan or MRI to check the status of the disease.
- Blood (about 5-6 teaspoons) will be drawn for routine tests, biomarker testing (including genetic biomarkers), and to check for hepatitis B and C and HIV.
   Biomarkers are found in the blood/tissue and may be related to your reaction to the study drugs.
- You will have a tuberculosis (TB) skin test. For this test, fluid will be injected under the skin on your forearm, making a bump. Two (2) days later, you will return to the clinic to have the skin test checked. If you have ever been exposed to TB, the bump will still be there.
- Urine will be collected for routine tests.

- You will have a core biopsy for biomarker testing, which may include genetic biomarkers. To perform a core biopsy, a sample of tissue is removed using a hollow core needle that has a cutting edge.
- If you can become pregnant, within 7 days before your first dose of study drugs, blood (about ½ teaspoon) will be drawn for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other treatment options will be discussed with you.

## **Study Groups**

If you are found to be eligible to take part in this study, you will be assigned to a dose level of selumetinib based on when you join this study. Up to 40 participants will be enrolled in this study. All will take part at MD Anderson.

Up to 3 dose levels of selumetinib will be tested. Up to 3 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of selumetinib is found.

All participants will receive the same dose of tremelimumab and durvalumab.

If you were enrolled to receive the first 2 dose levels of selumetinib and the third dose level is found to be safe and tolerable, your dose may be increased to the third dose level. This will be discussed with you.

## **Study Drug Administration**

Each study cycle is 28 days.

You will be randomly assigned (as in the flip of a coin) to 1 of 2 study cohorts (groups). This is done because no one knows if one study group is better, the same, or worse than the other group. You will have an equal chance (50/50) of being assigned to either cohort:

- If you are in **Cohort 1**, you will take selumetinib on an intermittent schedule (alternating 7 days on, 7 days off). This means you will take selumetinib on Days 1-7 and Days 15-21 of each cycle. You will <u>not</u> take the study drug on Days 8-14 and 22-28.
- If you are in **Cohort 2**, you will take selumetinib every day.

You will take selumetinib 2 times every day. Each dose should be taken about 12 hours apart. You must fast (having nothing to eat or drink except water) for 1 hour before and F2 hours after taking selumetinib.

You should record each selumetinib dose in the dosing diary that will be given to you. You should bring the diary to your study visits at the end of every cycle.

You will also receive tremelimumab and durvalumab by vein over about 60 minutes each for each infusion on Day 1 of each cycle. After Cycle 4, you will only receive durvalumab. You will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

#### **Study Visits**

## About 14 days before the first dose of the study drugs:

- You will have a physical exam.
- Blood (about 3 teaspoons) will be drawn for routine tests.
- If the doctor thinks it is needed, you will have an EKG.

#### On Day 1 of each cycle:

- You will have a physical exam.
- Blood (about 3 teaspoons) and urine will be collected for routine tests.
- During Cycle 2, blood (about 5 teaspoons) will be drawn for biomarker testing, including genetic biomarkers.
- If the doctor thinks it is needed, you will have an eye exam.
- If you can become pregnant and the doctor thinks it is needed, blood (about ½ teaspoon) will be drawn for a pregnancy test.

On **Day 1 of Cycles 1 and 4** (about Week 16), you will have an EKG. During Cycle 1, you will have an EKG before and up to 3 hours after your dose of study drugs.

During **even-numbered cycles** (Cycles 2, 4, 6, and so on), you will have a CT scan or MRI to check the status of the disease.

**Every 3 cycles** starting with Cycle 3 (Cycles 6, 9, and so on), you will have an ECHO or MUGA scan.

**At any time while on study,** if the doctor thinks it is needed, the above tests/procedures (routine blood and urine collections and EKGs, for example) may be repeated.

## **Follow-Up Visits**

## At about 30 days and 90 days after your last dose of the study drugs:

- You will have a physical exam.
- Blood (about 3 teaspoons) will be drawn for routine tests.
- You will have an EKG.
- At the 90-day follow-up visit, blood (about 5 teaspoons) will be drawn for biomarker testing, including genetic biomarkers.
- If you can become pregnant and the doctor thinks it is needed, blood (about ½ teaspoon) will be drawn for a pregnancy test.

**About 60 days** after your last dose of study drugs, blood (about 3 teaspoons) will be drawn for routine tests.

If you stop taking the study drugs for any reason other than the disease getting worse, you will continue to have an MRI or CT scan to check the status of the disease about every 8 weeks. If the disease worsens, these scans will stop.

## Long-Term Follow-Up

Every 6 months for up to 2 years, the study staff will call you to ask how you are doing. These calls should last about 5-10 minutes.

## **Other Information**

- While taking selumetinib, avoid having any grapefruit, Seville (sour) oranges, star fruit, pomegranate, and products containing juices of these fruits.
- You should not donate blood after receiving selumetinib or durvalumab and for at least 12 weeks after receiving the last dose of the study drugs.
- You should avoid excessive exposure to sunlight.
- You should not take any vitamin E supplements while on study.
- You should pay attention to your oral care. While taking the study drug, you
  may develop dry lips or sores in your mouth that require additional care. This
  will be discussed with you.
- Ask the study doctor before taking any new drugs during the study. This
  includes over-the-counter drugs and herbal and natural remedies. You should
  avoid medications that may affect your liver. Your study doctor will review all of
  the drugs you are taking and let you know if they can be taken during the
  study.
- You should not receive any live vaccines (vaccines containing live organisms)
  from between 30 days of receiving durvalumab and 30 days after the last dose
  of durvalumab. The study doctor will discuss this with you in more detail. If you
  need a vaccine while on study, talk with the study staff before receiving it.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

Durvalumab, tremelimumab, and selumetinib may each cause low blood cell counts (red blood cells, platelets, and white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia, urinary tract infection, oral/dental infections, and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

## **Durvalumab Side Effects**

The study drug durvalumab works by boosting the immune system. Side effects as a result of stimulating the immune system have been reported in patients being given durvalumab. These immune system side effects are included in the risks outlined below. Durvalumab may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue.

## Common (occurring in more than 20% of patients)

| <ul><li>fatigue</li></ul> | <ul><li>dry/itchy skin</li></ul> | <ul> <li>loss of appetite</li> </ul> |
|---|---|---|
| <ul><li>skin rash</li></ul> | <ul><li>nausea</li></ul> | |

## Occasional (occurring in 3-20% of patients)

| <ul> <li>fever</li> <li>underactive thyroid</li> <li>overactive thyroid</li> <li>gland (possible</li> </ul> | <ul><li>pain (joint/muscle)</li><li>numbness/tingling</li></ul> |
|---|---|
| gland (possible weight gain, heart failure, and/or constipation) • vomiting • diarrhea • abnormal liver tests (possible liver damage) | <ul> <li>(hands/feet)</li> <li>abnormal kidney test<br/>(possible kidney<br/>damage)</li> <li>difficulty breathing</li> <li>cough</li> </ul> |

## Rare but serious (occurring in fewer than 3% of patients)

- heart inflammation
  immune system damage to the nervous system (causing numbness and/or paralysis)
- decreased production of adrenal hormones (possible weakness
- type 1 diabetes, which requires insulin
- high blood sugar
- inflammation of the intestines
- hole in the intestines (possibly leaking
- kidney inflammation (possible decreased kidney function)
- lung inflammation (possible difficulty breathing)
- allergic reaction

| and/or | low | blood |
|--------|------|-------|
| pressu | ıre) | |

- pituitary gland failure/inflammation (possible headaches, thirst, and/or irregular periods in women)
- contents into the abdomen)
- inflammation of the pancreas (possible abdominal pain)
- digestive system bleeding
- liver damage

 infusion reaction (possible chills, fever, difficulty breathing, and/or change in blood pressure)

## **Tremelimumab Side Effects**

The study drug tremelimumab works by boosting the immune system. Side effects as a result of stimulating the immune system have been reported in patients being given tremelimumab. These immune system side effects are included in the risks outlined below. Tremelimumab may cause unknown side effects resulting from your immune system attacking your organs. This may cause inflammation and inflammation-related side effects in any organ or tissue.

## Common (occurring in more than 20% of patients)

- fatigue (lack of energy)
- dry/itchy skin
- skin rash
- diarrhea

- nausea/vomiting
- loss of appetite

## Occasional (occurring in 3-20% of patients)

- fever
- headache
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)
- high blood sugar (possible diabetes)
- weight loss
- constipation
- dehydration
- inflammation of the intestines
- abdominal pain
- abnormal digestive blood test (possible inflammation of the pancreas)
- low red blood cell counts

- abnormal liver tests (possible liver damage)
- numbness/tingling (hands/feet)
- kidney inflammation (possible decreased kidney function)
- abnormal kidney test (possible kidney damage)
- difficulty breathing
- cough

# Rare but serious (occurring in fewer than 3% of patients)

- blood vessel inflammation (possible bleeding and/or bruising)
- pituitary gland failure/inflammation (possible headaches, thirst,
- lung inflammation or fluid build up in the lungs (possible difficulty breathing)

- inflammation of the arteries around the temples (possible pain and/or double vision)
- immune system damage to the nervous system (causing numbness, confusion, and/or paralysis)
- overactive thyroid gland (possible weight loss, heart rate changes, and/or sweating)
- decreased production of adrenal hormones (possible weakness and/or low blood pressure)

- and/or irregular periods in women)
- Type 1 diabetes
- inflammation of the pancreas (possible abdominal pain)
- holes in the intestines (possibly leaking contents into the abdomen)
- digestive system bleeding
- low blood cell counts (white/platelet)
- liver damage (hepatitis)

- weakness (arms/legs/face)
- allergic reaction
- infusion reaction (possible chills, fever, difficulty breathing, and/or change in blood pressure)
- immune system disease (possible dry mouth/eyes, joint pain, fatigue, and/or organ damage)

## **Selumetinib Side Effects**

## Common (occurring in more than 20% of patients)

skin rash (possibly acne-like)
 abnormal liver tests (possible liver damage)

## Occasional (occurring in 3-20% of patients)

- swelling (face)
- high blood pressure
- fever
- dizziness
- headache
- depression
- hair loss (partial or total)
- dry/itchy skin
- nail changes

- high blood levels of phosphate (possible kidney damage)
- low blood levels of potassium (possible weakness and/or muscle cramps)
- abdominal pain/swelling
- constipation
- dry mouth

- mouth blisters/sores (pain and/or difficulty swallowing)
- loss of appetite
- low blood cell count (red/platelets/white)
- pain (joint/back)
- blurred vision
- cough
- difficulty breathing

# Rare but serious (occurring in fewer than 3% of patients)

- severe heart problems
- heart failure

- hole in the intestines (possibly leaking contents into the abdomen)
- liver/kidney failure
- vision problems
- blood clot inside the eye (possible blindness)

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

## **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

**EKGs and ECHOs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

**MUGA scans** may cause allergic reactions to the radioactive tracer, injection site soreness, and/or swelling. They may cause damage to cells or tissue from being exposed to the radiation used in the scan. These side effects may occur in less than 10% of patients.

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the aspiration. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**Fasting** may cause your blood sugar to drop. You may feel tired, hungry, and/or nauseous. If you have diabetes, it is important to talk to your doctor about managing your blood sugar while fasting.

During the **eye exam**, your pupils will be dilated with eye drops to allow a good view of the back of the eye. This will result in some blurred vision lasting for a few hours. You will not be able to drive during this time.

During an **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

CT scans send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

The type of **genetic testing** being performed in this study will not provide you or your doctor information about diseases that are passed down in families. It will not tell the study researchers anything that will prevent you from getting health insurance, and it will not tell the study researchers anything about any diseases or conditions you may get in the future.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study. To protect your identity, the data and samples collected from you will be labeled with a unique number instead of your name or other identifying information. Only the study doctor or study staff will have access to the code that can link you to your data and samples.

This study may involve unpredictable risks to the participants.

## **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study and for at least 180 days after your last dose of selumetinib, durvalumab, and tremelimumab or 90 days after your last dose of selumetinib and durvalumab (whichever is the longer period), if you are sexually active.

Birth Control Specifications: You must use effective methods of birth control while on study. Effective methods include:

- barrier method or intrauterine device (IUD)
- hormonal methods (implants, patch, pill, mini-pill, and/or injections)

Talk with the study staff about which methods of birth control are acceptable to use.

Males: Do not donate sperm while on study and for at least 180 days after your last dose of selumetinib, durvalumab, and tremelimumab or 90 days after your last dose of selumetinib and durvalumab (whichever is the longer period). If your partner/spouse becomes pregnant while you are on this study, the sponsor would like to collect information about the pregnancy. The study sponsor's contact information will be made available so that, if you and your partner wish to, you can share information

about the outcome of the pregnancy with the sponsor. If you and/or your partner choose not to share this information, it will not result in any penalty or loss of benefits to which you are otherwise entitled.

Females: If you are pregnant or breast feeding a baby, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away. The sponsor will ask for information about the pregnancy.

Getting pregnant will result in your removal from this study.

#### OPTIONAL PROCEDURES FOR THE STUDY

**Optional Procedure #1:** If you agree, you will have a tissue biopsy on Day 21 of Cycle 1 for biomarker testing, including genetic biomarkers. To collect a tissue biopsy, the affected area is numbed with anesthetic and a small amount of tissue is removed using a large needle.

You do not have to agree to the optional procedures in order to take part in this study. There are no benefits to you for taking part in the optional procedure. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedure.

## **Optional Procedure Risks:**

Having **biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**Genetic research** may result in the development of beneficial treatments, devices, new drugs, or patentable procedures. There are no plans to provide you compensation from such developments. The results of any genetic tests may be put in your health records. If this information were released, it could be misused. Such misuse could be distressing, and it could cause you or your family members to have difficulty obtaining insurance coverage and/or a job.

#### CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES

Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have an additional biopsy on Day 21 of Cycle 1 for biomarker testing?

YES NO

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson, AstraZeneca, or MedImmune for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

#### **Additional Information**

- 4. You may ask the study chair (Dr. Don L. Gibbons, at 713-792-6363) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can then decide if you need to have any visits or tests to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, AstraZeneca, MedImmune, the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson. Possible reasons your participation may be stopped include if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.
- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is sponsored and/or supported by: AstraZeneca and MedImmune.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

Your personal information and/or samples are being collected as part of this study. These data and/or samples may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples or data at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

Before being shared for future research, every effort will be made to remove your identifying information from any data and/or samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or samples are used for future research. If this research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### **Genetic Research**

Samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

## **Conflict of Interest**

Outside relationships are disclosed to and approved by the Conflict of Interest Committee, which reviews these relationships for compliance with institutional policy. This review helps the IRB to assure that financial relationships do not have an impact on the conduct of this study. The following members of the study staff have disclosed compensation from the funding source(s) of this study:

John Heymach (Study Co-Chair)

#### <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and

study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:

- Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
- The IRB and officials of MD Anderson
- AstraZeneca and MedImmune, who are sponsors or supporters of this study, and/or any future sponsors/supporters of the study
- Any future sponsors and/or licensees of the study technology.
- Study monitors and auditors who verify the accuracy of the information
- Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the

| consent form for this study, or have had it read to me. I have had a cabout it, ask questions, and talk about it with others as needed. I giv | |
|---|---|
| permission to enroll me on this study. By signing this consent form, | _ |
| any of my legal rights. I will be given a signed copy of this consent of | document. |
| OLONIA TUDE: OF DADTIOIDANT | DATE |
| SIGNATURE OF PARTICIPANT | DATE |
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT | |
| I was present during the explanation of the research to be performed | d under this protocol. |
| | · |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT | DATE |
| PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) | |
| A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | |
| oner term series in present (TTT e) and patients time are limited. | |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT | |
| I have discussed this research study with the participant and/or his or<br>representative, using language that is understandable and appropria | |
| have fully informed this participant of the nature of this study and its | |
| and risks and that the participant understood this explanation. | possible solitonic |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |

Protocol 2017-0888 October 03, 2023 Page 17 of 17

| <u>TRANSLATOR</u> | | |
|---|---|---|
| I have translated the above informed consent as written (without additions or subtractions) into and assisted the people | | |
| Obtaining and providing consert consent process for this partici | nt by translating all questions and respon | nses during the |
| NAME OF TRANSLATOR | SIGNATURE OF TRANSLATOR | DATE |
| | nslator was a member of the research to<br>the translator, must sign the witness lin | • |